CLINICAL TRIAL: NCT02011724
Title: An Open Label, Multi Center, Post Marketing Study Of Pain And Quality Of Life Outcomes In Subjects With a Single Painful Venous Leg Ulcer Treated With Apligraf®
Brief Title: A Study Of Pain And Quality Of Life Outcomes In Subjects With a Single Painful Venous Leg Ulcer Treated With Apligraf®
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-VLU-003-AG
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Venous Leg Ulcers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apligraf (Experimental)
  Interventions: Device: Apligraf

INTERVENTIONS:
Device: Apligraf

SUMMARY:
The objective of the study is to demonstrate that treatment with Apligraf reduces venous leg ulcer (VLU)-related pain and improves the quality of life (QOL) of patients with a painful VLU.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a minimum of 18 years of age.
* Subject has read, understood, and signed an Institutional Review Board (IRB)-approved Informed Consent Form (ICF).
* Subject is able and willing to follow study procedures and instructions.
* Subject reports moderate VLU-related pain (defined as ≥4 based on maximum pain level over preceding 24 hours) on numeric rating scale (NRS) at both Week -2 and Day 0).
* Subject has a partial or full-thickness VLU between 1-60 cm2 and 1-36 months duration, which, in the opinion of the Investigator, has not adequately responded to conventional ulcer therapy.
* Female subject of childbearing potential has a documented negative urine pregnancy test.
* Subject (male or female) agrees to use highly effective methods of contraception for the duration of the study.

Exclusion Criteria:

* Subject has more than 1 VLU.
* Female subject who is lactating.
* Subject with significant or severe non VLU-related chronic pain which, in the Investigator's opinion, would impact subject's ability to evaluate their VLU-related pain. Subject with non-VLU-related chronic pain must be on a stable pain medication regimen and must, in the Investigator's opinion, not be anticipated to require a new pain medication for the chronic pain condition during the course of the study.
* Subject is not willing to discontinue the use of topical analgesics at the VLU (topical anesthetic is permitted for debridement).
* Subject who has arterial disease, as determined by an ankle-brachial index (ABI), of <0.65.
* Subject who has received an investigational drug, device, or biological/bioactive treatment within 30 days prior to study enrollment.
* Subject who is scheduled to have a vascular intervention on the study extremity during the study.
* Subject with a biopsy confirmed active malignancy at the VLU. Also, subject with any active malignancy not at the VLU, with the exception of squamous cell carcinoma or basal cell carcinoma.
* Subject who is currently receiving, anticipates receiving, or has received, at any time within 30 days prior to Screening visit, topical corticosteroids at the VLU.
* Subject has vasculitis, severe rheumatoid arthritis, and other collagen vascular diseases.
* Subject has signs and symptoms of wound infection, cellulitis, or osteomyelitis at the VLU.
* Subject has a VLU with an avascular wound bed.
* Subject has a VLU with exposed bone, tendon, or fascia.
* Subject has other wounds (DFU, surgical, etc.) on the same limb as the VLU.
* Subject has a known hypersensitivity to bovine collagen or to the components of the Apligraf agarose shipping medium.
* Subject previously treated with Apligraf, or any other cell or tissue-based product at the VLU within 30 days of the Screening visit.
* Subject who, in the opinion of the Investigator, has a history of alcohol or substance abuse within the previous year that could interfere with study compliance (eg, inability to attend scheduled study visits).
* Subject, who in the opinion of the Investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Percent reduction in maximum VLU-related pain at Week 5 | Day 0 - Week 5
  Based on the maximum pain levels during the preceding 24 hours

SECONDARY OUTCOMES:
Reduction in maximum VLU-related pain at 48 hours following initial Apligraf application | Day 0 - 48 hours after Apligraf application
Reduction on SF-12v2 - Pain Enhanced Health Survey at Week 5 | Day 0 - Week 5
Reduction in class and/or dose of VLU-related pain medications at Week 5 | Day 0 - Week 5
Reduction on Cardiff Wound Impact Schedule (CWIS) at Week 5 | Day 0 - Week 5

OTHER OUTCOMES:
Reduction in average VLU-related pain at Week 5. | Day 0 - Week 5
Reduction in VLU-related pain using both maximum and average pain | Day 0 - Weeks 1, 2, 3, and 4
  From baseline (Day 0) to Weeks 1, 2, 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: William A. Marston, MD, Principal Investigator — Division of Vascular Surgery, UNC at Chapel Hill; Scott Gorenstein, MD, Principal Investigator — Winthrop University Hospital; David G. Armstrong, DPM, MD, PhD, Principal Investigator — Department of Surgery, University of Arizona College of Medicine
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States